CLINICAL TRIAL: NCT06905613
Title: Technical Feasibility Study of a Novel Wearable Capnograph (MARIE) in an Emergency Care Environment, Part 1
Acronym: MARIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Oxlantic Medical AB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5.1-2024-76464
Record Dates: First submitted 2024-12-16; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Technical Feasibility; Ambulances
Keywords: MARIE Capnograph; MARIE Nasal Adapter Set O2 - Adult; Mainstream Respiratory Infrared Equipment; capnograph

STUDY DESIGN:
Intervention Model Description: In the first step we will include 20 Healthy volunters and if no AE we plan to include 30 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Technical feasibility study of a novel wearable capnograph (MARIE) in an emergency care environmen (Other): MARIE will be connected to the patient by attaching the nasal adapter set and connecting the CO2 sensor. ETCO2 and RR values will be logged before and during the transport by writing down the values in the Case Report Form (CRF). On arrival at the hospital ETCO2 and RR will be measured by a reference instrument and logged in to the CRF. There will be trained study personnel responsible for operating the investigational device and populating the CRF, capturing all information which is required according to the study protocol.
  Interventions: Device: Technical feasibility study of a novel wearable capnograph (MARIE) in an emergency care environment

INTERVENTIONS:
Device: Technical feasibility study of a novel wearable capnograph (MARIE) in an emergency care environment — MARIE will be connected to the patient by attaching the nasal adapter set and connecting the CO2 sensor. ETCO2 and RR values will be logged before and during the transport by writing down the values in the Case Report Form (CRF). On arrival at the hospital ETCO2 and RR will be measured by a reference instrument and logged in to the CRF. There will be trained study personnel responsible for operating the investigational device and populating the CRF, capturing all information which is required according to the study protocol.
  Other Names: Capnograph; MARIE

SUMMARY:
You have been assessed by paramedics as needing to go to the emergency department. During transport, the paramedics will monitor you by, for example, measuring your blood pressure and checking your pulse.

In healthcare, we are constantly working to improve and optimize the degree of monitoring during ambulance transports and through this also be able to start adequate treatment earlier. In this case, we are working to understand whether exhaled carbon dioxide levels can be used to monitor important processes in the body during ambulance transport. Therefore, we offer you to participate in a project that deals with whether we can use a new equipment to measure and monitor exhaled carbon dioxide during the journey to hospital.

This clinical trial is being conducted in Region Uppsala in collaboration with Oxlantic Medical AB. The main responsible and Sponsor for the trial is Oxlantic Medical AB. The research lead for the trial is Region Uppsala and Uppsala University.

This clinical trial has been subject to ethical review and approved by the Ethics Review Authority.

ELIGIBILITY:
Inclusion Criteria:

* 20 healthy volunteers 18-84 years
* 30 patients between 18-84 years being transported by ambulance

Exclusion Criteria:

* Priority 1 ambulance transports
* Patients needing oxygen supply
* Known pregnancy
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Adequate values of ETCO2 and respiratory rate | During ambulance transport from the start of the transport to the arrival at the emergency department
  Verifying that credible measurements of EtCO2 and Respiratory Rate are reported during the transport.

CONTACTS AND LOCATIONS:
Overall Officials: David Smekal, MD, PhD, docent, Principal Investigator — Department of Surgical Sciences
Locations (1):
- Ambulansstationen Uppsala Region, Uppsala, Uppsala County, Sweden